CLINICAL TRIAL: NCT04838483
Title: Clinical Performance of Indirect Adhesive Restorations Luted With Light-cured Composite Resin
Brief Title: Clinical Performance of Posterior Indirect Adhesive Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gulsah YENIER, Assist.Prof., Okan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2/25
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Dental Caries; Endodontically Treated Teeth; Dental Restoration Failure of Marginal Integrity; Wear, Occlusal
Keywords: Indirect restoration; Adhesive restoration; Cementation; Composite resin
MeSH Terms: conditions — Dental Caries; Tooth, Nonvital; Tooth Attrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indirect restorations luted with light-cured composite resin. (Experimental): Subjects for the study will be identified from patients who had treated with indirect adhesive restorations onlay or overlay during the period 2016 to 2017 was performed at Istanbul Okan University Faculty of Dentistry by an experienced clinician.
  Local anesthesia was applied if necessary. After caries and/or failed restorations were removed, the preparations were performed according to defined principles for adhesive onlays/overlays. At least one cuspal coverage was required for each restoration. All undercuts were eliminated using composite resin. Following the cavity preparation, immediate dentin sealing was applied and polymerized prior to impression taking. Indirect restorations were designed and fabricated with CEREC system. Surface treatments and clinical protocols were performed under manufacturer's instructions. Adhesive cementation with composite resin procedure was carried out with the rubber-dam isolation.
  Interventions: Device: Indirect adhesive restoration of posterior teeth

INTERVENTIONS:
Device: Indirect adhesive restoration of posterior teeth — Indirect restoration of significant loss of dental hard tissue
  Other Names: Ceramic onlay or overlay

SUMMARY:
Clinical performance of indirect adhesive restorations - onlays, overlays- luted with light-cured composite resin will be evaluated.

DETAILED DESCRIPTION:
Indirect adhesive restorations are indicated in large Class II defects, replacement of large compromised existing restorations or endodontically treated teeth where cuspal protection is required. The need to perform adhesive restorations of posterior teeth is not only linked to esthetic purposes, but also have possibility of strengthening the remaining tooth structure. Indirect technique decreases polymerization shrinkage, reduces microleakage and also improves the marginal seal when comparing direct resin composites. Furthermore, it provides improved physical and mechanical properties, ideal occlusal morphology, more precise control of proximal contours and contacts. Indirect adhesive restorations are classically delivered with an adhesive procedure including dual-cure cement. Updated approaches now include the use of composite resins as luting agent.

This study will be carried out as a prospective study, with assessment of the restorations after three years. PASS 11 Software was used to calculate the sample size. At least 77 indirect adhesive restorations will be included for this study. Patients referred to Istanbul Okan University Faculty of Dentistry between 2016-2017 who had returned for the baseline recall and at least one year recall after the treatment will be invited for eligibility to participate in the study. 83 indirect adhesive restorations in at least 60 patients will be included. The patients who will not meet all the inclusion criteria will be excluded from the study. A signed informed consent form will be obtained from all patients before beginning the study.

Restorations will be evaluated clinically according to FDI World Dental Federation criteria. Three main groups- esthetic, functional, biological properties- and their sub-categorizes of FDI World Dental Federation criteria will be scored on a scale of 1 to 5. Statistical analysis will be performed using R (v.3.5.3) Software and the SIGN.test function in the BSDA package (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Significant loss of dental hard tissue
* Endodontically treated teeth in posterior region
* Replacement of large compromised existing restoration
* Large Class II restoration
* Age of 18-60 years
* Good oral hygiene
* Presence of interproximal contact to at least one neighboring teeth • In occlusion with antagonist teeth
* Cavity preparation with at least one cuspal coverage

Exclusion Criteria:

* Serious medical problems or allergies to substances and/or products to be used
* Severe periodontal problems
* Poor oral hygiene
* Direct pulp capping
* Presence of parafunctional behaviors
* Pregnant or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Survival rate | at 5 years
  FDI World Dental Federation criteria functional properties

SECONDARY OUTCOMES:
Esthetic properties | at 5 years
  FDI World Dental Federation criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Yenier, DDS, PhD, Principal Investigator — Istanbul Okan University Faculty of Dentistry
Locations (1):
- Istanbul Okan University Faculty of Dentistry, Istanbul, Tuzla, Turkey (Türkiye)

REFERENCES:
- [Background] D'Arcangelo C, Zarow M, De Angelis F, Vadini M, Paolantonio M, Giannoni M, D'Amario M. Five-year retrospective clinical study of indirect composite restorations luted with a light-cured composite in posterior teeth. Clin Oral Investig. 2014;18(2):615-24. doi: 10.1007/s00784-013-1001-8. Epub 2013 May 22. PMID 23695612
- [Background] Veneziani M. Posterior indirect adhesive restorations: updated indications and the Morphology Driven Preparation Technique. Int J Esthet Dent. 2017;12(2):204-230. PMID 28653051
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Magne P, Razaghy M, Carvalho MA, Soares LM. Luting of inlays, onlays, and overlays with preheated restorative composite resin does not prevent seating accuracy. Int J Esthet Dent. 2018;13(3):318-332. PMID 30073216
- [Background] D'Arcangelo C, Vanini L, Casinelli M, Frascaria M, De Angelis F, Vadini M, D'Amario M. Adhesive Cementation of Indirect Composite Inlays and Onlays: A Literature Review. Compend Contin Educ Dent. 2015 Sep;36(8):570-7; quiz 578. PMID 26355440
- [Background] Naeselius K, Arnelund CF, Molin MK. Clinical evaluation of all-ceramic onlays: a 4-year retrospective study. Int J Prosthodont. 2008 Jan-Feb;21(1):40-4. PMID 18350945
- [Derived] Yurdaguven GY, Ciftcioglu E, Kazokoglu FS, Kayahan MB. 5-Year clinical performance of ceramic onlay and overlay restorations luted with light-cured composite resin. J Dent. 2024 Oct;149:105258. doi: 10.1016/j.jdent.2024.105258. Epub 2024 Jul 25. PMID 39067649